CLINICAL TRIAL: NCT02768948
Title: Telmisartan Promotes the Differentiation of Monocytes Into Macrophages M2 in Diabetic Nephropathy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-AOI-09
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telmisartan (Experimental): treatment with telmisartan at doses of 80 mg / day for 6 months
  Interventions: Drug: telmisartan during 6 months; Procedure: blood sample
- losartan (Experimental): Losartan at a dose of 100 mg / d for 6 months.
  Interventions: Drug: Losartan during 6 months; Procedure: blood sample

INTERVENTIONS:
Drug: telmisartan during 6 months — telmisartan during 6 months
  Arms: telmisartan
Drug: Losartan during 6 months — Losartan during 6 months
  Arms: losartan
Procedure: blood sample — blood sample

SUMMARY:
The severity of the diabetic nephropathy is proportional to proteinuria rate and degree of renal interstitial fibrosis. Despite many treatments available today, diabetic nephropathy is responsible for a quarter of cases of end-stage renal disease (ESRD) requiring the use of renal replacement therapy or kidney transplantation. It develops as follows: chronic hyperglycemia of diabetes abyss renal glomeruli that allow proteins in the urine room. In response, the tubular epithelium produces monocyte chemoattractant protein-1 (MCP-1) that attracts monocytes circulating in the renal interstitium. Monocytes then differentiate into M1 or M2 macrophages. M1 macrophages increased MCP-1 production while M2 macrophages produce transforming growth factor beta (TGF-β) pro-fibrogenic. Renal fibrosis is negatively correlated with the glomerular filtration rate itself proportional to the number of nephrons. The decrease in the number of nephrons majorises secondarily proteinuria by the onset of focal segmental glomerulosclerosis lesions. Production of MCP-1 increases with the renal proteinuria because M1 macrophages earning kidneys reinforce the production of MCP-1, and fibrosis worsens because M2 macrophages infiltrate in turn kidneys and produce TGF -β.

A way of limiting renal fibrosis would be to decrease renal monocytic infiltration by promoting the differentiation of monocytes towards macrophages M2. Although more numerous, M2 macrophages no longer benefit the kidneys because the decline of M1 macrophages decrease renal MCP-1 production. Ex vivo IL1-β orients the differentiation of monocytes towards macrophages M1 and IL-4 to M2. By cons in vivo, the differentiating factors are poorly known. It is remarkable that metformin and telmisartan increase M2 macrophages M1 macrophages and decrease, respectively, in humans and mice. Moreover, telmisartan reduces proteinuria more than losartan in diabetic nephropathy in humans and Metformin decreases the amount of TGF-β intra-renal mice. This effect of telmisartan is independent of the type 1 receptor of angiotensin II (AT1R) since it is not obtained with losartan.

Telmisartan is a partial agonist of peroxisome proliferator-activated receptor gamma (PPARgamma), the working assumption is that telmisartan fosters the transition of monocytes to macrophages M2 form, and limit the recruitment of more monocytes in the kidneys and therefore proteinuria and renal fibrosis. To show this, it will be compared the ability of monocytes to differentiate ex vivo in M1 or M2 macrophages in diabetic nephropathy patients treated with losartan or telmisartan then it will characterize the role of PPARgamma in the monocyte / macrophage transition. Finally, it will be compared the urinary excretion of amino terminal propeptide of procollagen type 3 (PIIINP), considered a marker of renal fibrosis in patients receiving losartan or telmisartan.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes ;
* Proteinuria ≥ 0.5 g / g motivating the prescription of ACE inhibitors or ARA2 full dose;
* Processing statin;
* Processing metformin;
* court treatment with GLP-1 agonists and DPP-4 inhibitor;
* About who signed the informed consent;
* affiliated to the social security issue

Exclusion Criteria:

* Diabetic nephropathy not;
* GFR <30 ml / min / 1.73 m2;
* Type 1 diabetes;
* Maturity Onset Diabetes of the Youth (MODY);
* Use of telmisartan in the 6 months prior to enrollment;
* Liver cirrhosis (potential production of PIIINP);
* chronic inflammatory disease;
* active cancer;
* immunosuppression;
* Pregnant or breastfeeding women (urine pregnancy test will be performed for women of childbearing age);
* adult person under guardianship;
* Hospitalized person without his consent and not protected by law; person deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2020-07-11 (Actual)

PRIMARY OUTCOMES:
number of differentiation marker | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No